CLINICAL TRIAL: NCT05029180
Title: International Termination of Resuscitation Practices - a Worldwide Survey
Brief Title: International Termination of Resuscitation Practices
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ulrik Havshøj, MD, PhD student, University of Southern Denmark
Other Study IDs: 20/55990
Record Dates: First submitted 2021-08-11; First posted 2021-08-31 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Termination of resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Termination of resuscitation — Do estimate the approaches used worldwide when terminating resuscitative efforts

SUMMARY:
Neither the international nor the interregional variation in survival following OHCA is fully understood, but may rely on multiple factors such as: organization of the Emergency Medical Service (EMS) system bystander cardiopulmonary resuscitation (CPR), the use of Automatic External Defibrillators (AED's), response time, and which subgroups are included as the denominator, (i.e. obvious dead, withholding of resuscitation). Variation in denominators provide an obstacle when comparing outcome between different EMS-systems. Studies have found that Utstein factors explained half of the variation in survival to hospital discharge among different EMS agencies highlighting the importance of further research.

Due to the high mortality rate of OHCA, the decision of withholding or withdrawing resuscitative efforts must be made frequently. We find that a description of the differences in initiation and termination of resuscitation of adult patients (>18 years of age), suffering from non-traumatic OHCA could add an important perspective on the impact of differences in EMS systems across the World regarding the outcome following OHCA.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is a leading cause of death in the World. Substantial international differences in survival to hospital discharge has been reported; ranging from 3.1% to 20.4% worldwide, 0% to 18% in Europe, 0,5% to 8,5% in Asia, 9% to 17% in Australia and New Zealand and from 1.1% to 8.4% in North America. Regional differences of up to a fivefold increase in survival have also been reported in multiple settings and geographic locations.

Neither the international nor the interregional variation is fully understood, but may rely on multiple factors such as: organization of the Emergency Medical Service (EMS) system bystander cardiopulmonary resuscitation (CPR), the use of Automatic External Defibrillators (AED's), response time, and which subgroups are included as the denominator, (i.e. obvious dead, withholding of resuscitation). Variation in denominators provide an obstacle when comparing outcome between different EMS-systems. Studies have found that Utstein factors explained half of the variation in survival to hospital discharge among different EMS agencies highlighting the importance of further research.

Due to the high mortality rate of OHCA, the decision of withholding or withdrawing resuscitative efforts must be made frequently. The European Resuscitation Council (ERC) stated in their 2021 guidelines that:

1. "Systems should implement criteria for the withholding and termination of CPR out-of-hospital cardiac arrest (OHCA), taking into consideration the specific local legal, organizational, and cultural context."
2. "Systems should define criteria for the withholding and termination of CPR, and ensure criteria are validated locally."
3. "Systems should implement criteria for early transport to hospital in cases of OHCA, taking into account the local context, if there are no criteria for withholding/terminating CPR".

To validate Termination of Resuscitation rules locally could be challenging both ethically and epidemiologically. This would require a prospective study with a transportation rate of 100%, which could put an immense amount of pressure on the limited sources of the EMS system, and moreover providing sufficient power in the study could be difficult.

We find that a description of the differences in initiation and termination of resuscitation of adult patients (>18 years of age), suffering from non-traumatic OHCA could add an important perspective on the impact of differences in EMS systems across the World regarding the outcome following OHCA.

ELIGIBILITY:
Inclusion Criteria:

* Countries that provide two separate answers

Exclusion Criteria:

* Countries that do not provide two separate answers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: International experts in OHCA
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-05-16 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in termination of resuscitation practices - a questionnaire | 1 year
  legislation, termination rules, cultural differences, regional differences, description

IPD SHARING:
Plan to Share IPD: No
There are no data regarding patients in this study

DOCUMENTS (1):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT05029180/Prot_000.pdf